CLINICAL TRIAL: NCT06521242
Title: The Effect of Training Given According to the Roy Adaptation Model on the Sleep and Quality of Life of Individuals With Hypertension
Brief Title: The Effect of Training Given to With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kader ÖZTÜRK (Other)
Responsible Party: Sponsor-Investigator, Kader ÖZTÜRK, Ass. Prof., Ataturk University
Organization: Ataturk University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Kader
Record Dates: First submitted 2024-06-26; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Hypertension; Train Sickness
Keywords: Nursing; Hypertension; Roy Adaptation Model; Sleep Quality; Quality of Life
MeSH Terms: conditions — Hypertension; Sleep Initiation and Maintenance Disorders | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Education (Experimental): The RAM-Based Training and Hypertension Training Manual were given to the intervention group for 8 weeks, once a week, for 2 hours each session. The patients in the intervention group were called during the 1st and 3rd weeks of the study, and telephone counseling was provided. Reminders were made for important points in RAM-based hypertension training in these meetings.
  Interventions: Other: Patient Education
- Control Group (No Intervention): Routine nursing care was given to the patients in this group without any training.

INTERVENTIONS:
Other: Patient Education — The intervention group was given 120 minutes of training.
  Arms: Patient Education

SUMMARY:
The study was conducted to examine the effects of the training given according to the Roy Adaptation Model on the sleep and quality of life of individuals with hypertension.

DETAILED DESCRIPTION:
Nurses have responsibilities in the treatment of hypertension, especially in controlling blood pressure and risk factors. Patient evaluation, diagnosis, follow-up, medication management, patient training, counseling, and clinical management of patients are among the responsibilities of nurses. It has been reported in previous studies that insufficient sleep duration and sleep apnea cause hypertension. Hypertension patients have been reported to have lower sleep quality scores when compared to individuals with normal blood pressure.

Training given by nurses on issues such as the importance of sleep, providing the necessary sleep time, and resting the individual can turn hypertension into a controllable disease. Previous studies reported that hypertension reduces the quality of life of individuals. Quality of life of hypertension patients is affected by factors such as age, gender, educational status, genetics, and the negative consequences of the disease. These negative consequences can be organ damage, side effects of drugs used, other diseases, obesity, and sexual dysfunctions. The negative psychological state of patients can affect blood pressure, quality of life, and sleep patterns negatively.

Nurses come to the forefront especially with their educational roles in preventive healthcare services, ensuring adaptation to disease and rehabilitation services. One of the most common models used to guide nursing practice and training is the Roy Adaptation Model (RAM) in nursing. Since RAM is functional in compliance with treatment and coping with chronic diseases, it is used as a conceptual model to construct and test nursing theories.

In a study that was conducted by Seah and Tham using RAM, it was reported that individuals adapted better to their disease in a changing environment in the treatment of bulimia nervosa. In the study of Afrasiabifar, Karimi, and Hassani, it was reported that patient training based on RAM strengthened the adjustment in the physiological state and self-concept areas of patients. It was found in another study that patients who received RAM training used effective coping mechanisms to adapt to various symptoms and responded more positively to treatment. In a study conducted by Lok et al., it was found that Cognitive Stimulation Therapy significantly increased the quality of life. Also, in another study that was conducted according to RAM, it was reported that web-based training increased the quality of life significantly in the physiological field.

There may be problems in compliance with the disease, symptoms, disease management, and treatment in hypertension patients. Patient training given by nurses is important in ensuring compliance with the disease, treatment, and care of hypertension patients. It is considered that the training based on RAM will be beneficial in the training to be given by nurses. Studies conducted in Turkey show that it is necessary to increase social awareness about hypertension and use model-based training by nurses who provide care. Because patient compliance is mainly focused on in patient training in the treatment process of hypertension and it is considered the most important variable in the treatment process. The present study was conducted to determine the effects of the training given according to RAM on sleep and quality of life in patients diagnosed with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with hypertension for at least 6 months
* Having applied to clinics for follow-ups
* Knowing the diagnosis and being able to express it verbally
* Not having a communication problem
* Being literate

Exclusion Criteria:

* Incomplete data form
* Leaving the study at any stage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
Pittsburg Sleep Quality Index (PSQI) | up to eight weeks
  The index was developed by Buysse et al. in 1989 to evaluate the sleep duration and intensity of individuals. The scale has 11 items and 7 sub-dimensions. These items are scored between 0-3. The scores that can be obtained from the scale range from "0" to "21" points. The Turkish validity and reliability of the scale was conducted by Ağargün et al. in 1996. A high total scale score indicates poor sleep quality. A reliable, valid, and standard measurement of sleep quality is made with PSQI. The Cronbach Alpha Internal Consistency Coefficient of the scale is 0.80.

SECONDARY OUTCOMES:
SF-36 Quality of Life Scale | up to eight weeks
  The scale, which is widely used in health-related quality-of-life studies, was developed by Ware and Sherbourne. A high score on the scale indicates a good quality of life. The scores that can be obtained from the sub-dimensions and the sum of the scale vary between 0-100. A score approaching zero indicates poor health and 100 indicates good health. The Turkish validity and reliability of the scale was conducted by Pınar in 1995.

CONTACTS AND LOCATIONS:
Locations (1):
- Turkey, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No